CLINICAL TRIAL: NCT07324070
Title: New Methods Electroconvulsive Therapy Augmentation
Brief Title: Electroconvulsive Therapy Augmented With Transcranial Magnetic Stimulation for Treatment Resistant Depression
Acronym: RMTSECT2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Daniel Divácký, MD, Charles University, Czech Republic
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 102/25 S-IV Grant AP
Record Dates: First submitted 2026-01-05; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Major Depressive Disorder (MDD); Treatment Resistant Depression (TRD)
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Blue group (Experimental): active group
  Interventions: Device: Electroconvulsive therapy; Device: Transcranial Magnetic Stimulation
- Red group (Sham Comparator)
  Interventions: Device: Electroconvulsive therapy

INTERVENTIONS:
Device: Electroconvulsive therapy — transcranial magnetic stimulation in intermitent theta burst stimulation protocol plus electroconvulsive therapy
Device: Transcranial Magnetic Stimulation — Transcranial magnetic stimulation, intermitent theta burst stimulation or sham TMS
  Arms: Blue group

SUMMARY:
The RTMSECT2 study was design to compare the application of electroconvulsive therapy augmented by transcranial magnetic stimulation. Subject will be compared both within groups and in group using psychometric scales and different deliver energy

DETAILED DESCRIPTION:
The study is monocentric, sham - controlled, randomized and triple blind (subjects, ECT and TMS practitioners, psychological assessment and outcome assessor). Subjects are randomized into two arms.

The primary objective is to determine whether TMS priming using the iTBS protocol prior to ECT results in a reduction of the seizure threshold. iTBS is administered with the shortest possible latency before the ECT procedure itself, ideally within two minutes of iTBS completion. The target site is the left DLPFC. The ECT dose is determined via a titration method to identify the lowest energy level required to elicit an epileptic seizure (seizure threshold). From the second session onwards, a stimulus intensity of 6 times the seizure threshold (6xST) is applied.

Delivered energy is measured in percentage for TMS and ECT of the maximum charge that the devices are able to administer. In the event of inadequate seizure duration, the dose will be increased by 100% at the subsequent session.

Primary outcome of the study is the overall apllied dose. Then Time to Recovery (TTR) is measured in minutes until fully awake. The subjects will be closely monitored throughout the entire ECT courses including psychometric scales.

The MECTA SIGMA device will be used for ECT. The Deymed DuoMAG XT will be used for TMS/iTBS.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to 18 or higher
* MADRS (Montgomery-Asberg Depression Scale) qual or higher than 20
* Major depressive disorder according to ICD 10

Exclusion Criteria:

* Other axis 1 disorder (for example schizofrenia, addiction, etc.)
* No dementia
* ECT in the last 3 months
* TMS in the last 3 months
* Psychotic disease or symptoms
* Ppregnancy or lactation
* Any neurological disease (for example epilepsy, etc.)
* Participation in another clinical trial within the last 30 days
* somatic condition which contraindicates ECT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2028-01-05 (Estimated); Study Completion 2029-01-05 (Estimated)

PRIMARY OUTCOMES:
reduction of the seizure treshold of ECT | during each ECT procedure
  determine whether TMS priming using the iTBS protocol prior to ECT results in a reduction of the seizure threshold

SECONDARY OUTCOMES:
Time to Recovery (TTR) | immediately after each ECT procedure
  The duration from ECT administration to the restoration of full consciousness, will be measured in minutes and assessed using a modified Glasgow Coma Scale.
speed of onset of antidepressant effect | T1: baseline and T2: during the course of ECT, between second and third ECT application (day 4)
  according to MADRS
MADRS response rate to treatment | T1: baseline, T2: during the course of ECT, between second and third ECT application (day 4), T3: after the course of ECT, within 2 days
  Percentage of participants experiencing a 50% decrease in MADRS
MADRS total response | T1: baseline, T2: during the course of ECT, between second and third ECT application (day 4), T3: after the course of ECT, within 2 days
  change in total MADRS score
AMI - SF (Autobiographical Memory Interview - short form) | T1: baseline, T3: after the course of ECT, within 2 days
  This scale is intended to quantify retrograde amnesia following electroconvulsive therapy (ECT).
QIDS (The Quick Inventory of Depressive Symptomatology) | T1: baseline, T2: during the course of ECT, between second and third ECT application (day 4), T3: after the course of ECT, within 2 days
  scale for self - assessment of depressive symptoms
ECCA (Electroconvulsive cognitive assesment) | T1: baseline, T2: during the course of ECT, between second and third ECT application (day 4), T3: after the course of ECT, within 2 days
  cognitive scale optimized for patients undergoing ECT
MoCA (Montreal Cognitive Assessment) | T1: baseline, T3: after the course of ECT, within 2 days
  screening test for cognitive functions, one of inclusion criteria of the study
TMT (trail making test) | T1: baseline, T3: after the course of ECT, within 2 days
  psychometric test for evaluation of cisual-perceptual and executive functions
RAVLT (The Rey Auditory Verbal Learning Test) | T1: baseline, T3: after the course of ECT, within 2 days
  Neuropsychological assessment designed to evaluate verbal memory in patients

CONTACTS AND LOCATIONS:
Locations (1):
- General University Hospital, Psychiatry department, Prague, Czech, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data can be shared when requested from a verified researcher
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available after the end of the study
Access Criteria: request by a verified researcher only